CLINICAL TRIAL: NCT04038593
Title: Feasibility and Effects of a Standardized Musical Intervention on Complex Dressing Care During Home Hospitalization: a Controlled and Randomized Study
Brief Title: Impacts of a Standardized Musical Intervention on Complex Dressing Care During Home Hospitalization (MUCAFOCSS)
Acronym: MUCAFOCSS
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID
Sponsor: Fondation Oeuvre de la Croix Saint-Simon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: FOCSS-2019-1; 2019-A01320-57 (Other: Agence Nationale de Sécurité du Médicament (ANSM) ID-RCB)
Record Dates: First submitted 2019-07-13; First posted 2019-07-31 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Bandage; Pain; Anxiety
Keywords: Pain; Anxiety; Complex dressing; Home hospitalization; Music
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Non interventional arm (No Intervention): Standard conditions of complex dressing cares, without experimental intervention. It will be a control intervention
- Comparative arm with relaxation music from Youtube© (Active Comparator): Standard conditions of complex dressing cares + use of non standardized music relaxation during complex dressing cares
  Interventions: Other: Youtube© relaxation music
- Interventional arm with MUSIC CARE© (Experimental): Standard conditions of complex dressing cares + administration of a specific music therapy program (U method) delivered through headphones from a tablet, under the direction of trained nurses.
  Interventions: Device: MUSIC CARE© intervention

INTERVENTIONS:
Other: Youtube© relaxation music — Use of non standardized relaxation music with Youtube© during cares
  Other Names: Youtube© condition
  Arms: Comparative arm with relaxation music from Youtube©
Device: MUSIC CARE© intervention — Use of MUSIC CARE© during cares
  Other Names: MUSIC CARE© condition
  Arms: Interventional arm with MUSIC CARE©

SUMMARY:
In France, home hospitalization services (HAD) are developing as an alternative to conventional hospitalization. In order to intervene at patients' home, a reason for referral must be defined. The most common one on the national territory is "complex dressing". Cares associated with these dressings can lead to symptoms such as pain and/or anxiety, and thus decrease the patient's quality of life. These two symptoms may be related, with the presence of one increasing the intensity of the other. Thus, drug treatments are often implemented as part of care, but may not be sufficient to relieve patients. Music has many interests in patients' pain and anxiety. MUSIC CARE© application allows the implementation of standardized musical interventions. It has been shown to be effective in reducing acute and chronic pain and anxiety in many clinical settings.

The aim of this study is to evaluate the feasibility of implementing MUSIC CARE© in the care of complex dressings at home and to confirm its effectiveness on the symptoms experienced by patients. In addition, attention will be paid to the impact of this standardized musical intervention on care time, medication use during care and patients' and caregivers' satisfaction.

DETAILED DESCRIPTION:
Complex dressing reason for referral represent one of the most frequent case in home hospitalization (HAD) referrals, accounting for 28.4% of HAD days in 2018 at national level. They can occur for different pathologies. They involve daily or several times a week care to repair dressings, monitor wound progress and healing.

Complex dressings care can lead to symptoms for the patient such as pain and/or anxiety. Those symptoms can be related. In fact, anxiety could influence the patient's feelings and assessment of pain.

MUSIC CARE© allows the implementation of standardized musical interventions. This technique can be compared to sophrology and hypnosis, but verbal suggestions are replaced by musical suggestions. This application is considered effective in reducing acute and chronic pain, reducing anxiety, reducing drug use in different clinical settings, and developing good patient satisfaction by international literature.

The hypothesis of this study is that the use of MUSIC CARE© during complex dressing home care could reduce patients' pain and anxiety, reduce patients' requests for drug treatments, reduce the time required for care, and develop a positive level of satisfaction among patients and caregivers.

Participants will be recruited during their hospitalization at the HAD of Fondation Oeuvre de la Croix Saint-Simon (Ile de France). A randomization list will be created upfront to determine the order of passage under the experimental conditions. After verification of the inclusion criteria and study proposal, patients who agree to participate will sign a free and informed consent form and will be assigned a coded identification number. They will respond to two measurement times, one before and one after the care. Caregivers will also complete questionnaires In order to obtain statistically exploitable results, 250 patients will be included.

ELIGIBILITY:
Inclusion Criteria:

* reason for referral "complex dressing"
* age > 18 year old
* inform consent
* pain numerical scale ≥3 during care
* able to speak and write French

Exclusion Criteria:

* patients with a deficiency in auditive function
* patients diagnosed with psychiatric pathologies
* so-called vulnerable patients, ie under guardianship or curatorship, or deprived of their liberty by a judicial or administrative decision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-01 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Pain felt during the care: numerical scale | Immediately after the intervention
  Measurement by a numerical scale (0 the minimum to 10 the maximum)

SECONDARY OUTCOMES:
Anxiety measurement | Immediately before/after the intervention
  Measurement assessed by numerical scale (0 the minimum to 10 the maximum)
Time needed for the care | Immediately before/after the intervention
  Measurement by caregivers
Satisfaction of patient and caregivers: numerical scale | Immediately after the intervention
  Measurement by numerical scale (0 the minimum to 10 the maximum)
Treatment request by the patient during the care | Immediately after the intervention
  Measurement by a dichotomous question (Yes/No)

CONTACTS AND LOCATIONS:
Overall Officials: Jérémy Martin, Principal Investigator — Fondation Oeuvre de la Croix Saint-Simon
Locations (1):
- Fondation Oeuvre de la Croix Saint-Simon, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No